CLINICAL TRIAL: NCT00035685
Title: Exposure of Children With Asthma to Household Environmental Tobacco Smoke
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 998; R01HL068828 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To examine whether or not primary school-aged children with asthma from low-income households have lower household environmental tobacco smoke (ETS) exposure than matched control children.

DETAILED DESCRIPTION:
BACKGROUND:

Children with asthma are particularly vulnerable to environmental tobacco smoke (ETS). However, despite this special vulnerability to ETS, children with asthma are at least as likely to live in smoking households, as are healthy children. Controversy exists, however, about whether or not the smoking members of households with children with asthma use specific strategies to reduce the harmful effects of their smoking on their children more than the smoking members of households of healthy children.

DESIGN NARRATIVE:

The case-control study examines whether or not primary school-aged children with asthma from low-income households have lower household ETS exposure than matched control children. Household ETS exposure will be measured by both objective monitoring, specifically passive nicotine dosimeters and child cotinine assays (the primary hypothesis), and maternal-report (the secondary hypothesis). Ninety children with physician diagnosed asthma and smoking mothers will be matched by age, gender, race/ethnicity, and other relevant variables to 90 healthy children. All children will be recruited from Metro Denver clinics providing services to low-income, underserved populations. The sample will contain equal numbers of African Americans, Hispanics, and Whites. Recruitment will target low-income populations due to their increased prevalence of, and associated morbidity from both asthma and tobacco smoking. Specific household smoking behaviors, as reported by mothers, will be examined for association with household nicotine and child cotinine levels. Finally, a set of carefully chosen measures will be examined in tertiary, exploratory analyses to help understand, clarify, and contextualize the observed results.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2001-12; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Walboldt — National Jewish Medical & Research Center